CLINICAL TRIAL: NCT02599688
Title: An Open-label Extension Study of the Safety and Efficacy of Subconjunctival Liposomal Latanoprost (POLAT-001) in Patients With Ocular Hypertension and Primary Open Angle Glaucoma
Brief Title: Open Label Extension of LipoLat-CS202
Status: Completed | Type: Observational
Sponsor: Peregrine Ophthalmic (Industry)
Responsible Party: Sponsor
Other Study IDs: LipoLat-CS203
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Results first posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Observation only — No intervention in this study.

SUMMARY:
This is an open-label, observational extension of patients who received POLAT-001 in LipoLat-CS202.

ELIGIBILITY:
* Inclusion criteria

  1. Successful completion of 3 months of participation in Study LipoLat-CS202.
  2. Treatment with POLAT-001 in Study LipoLat-CS202.
  3. Able and willing to give signed informed consent and follow study instructions.
* Exclusion criteria

Excluded from the study will be individuals with the following characteristics:

1. The development, during study LipoLat-CS202, of any exclusion criteria from that study (e.g., concomitant medication or co-morbid disease).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were randomized to received POLAT-001 and successfully completed LipoLat-CS202
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Professional Research Network, Goose Creek, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Post Treatment Follow-up: Post treatment follow-up
Period: Overall Study
Arm/Group | Post Treatment Follow-up
Started | 18
Completed | 14
Not Completed | 4
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1
Not completed — Termination by Sponsor | 2

BASELINE CHARACTERISTICS:
Arm/Group | Post Treatment Follow-up
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (7.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Description: Mean change from baseline (Visit 1 in Study LipoLat-CS202, NCT02466399) IOP at Month 3 (6 months after treatment in LipoLat-CS202).
Time Frame: 3 months
Population: Per protocol
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Post Treatment Follow-up
Number analyzed (Participants) | 16
mm Hg | -4.2 (4.0)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Post Treatment Follow-up
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 16/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Post Treatment Follow-up (N=18)
Infections and infestations (Infections and infestations) | 5 (7)
Musculoskeletal and connective tissue disorders (Eye disorders) | 2 (3)
Conjunctival haemorrhage (Eye disorders) | 5 (5)
Conjunctival hyperaemia (Eye disorders) | 3 (3)
Foreign body sensation in eyes (Eye disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If multi-center study publication not published within two (2) years after the completion of the Study at all sites, Investigator may publish the results of the Study obtained by Investigator with 60 days notice to Sponsor